CLINICAL TRIAL: NCT03104777
Title: A Cluster Randomised Controlled Trial Using Behavioural Insights to Improve the Healthiness of Packed Lunches in Primary Schools in Derby
Brief Title: A Trial to Improve the Healthiness of Packed Lunches in Primary School Aged Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Public Health England (Other Government)
Collaborators: Derby City Council (Unknown); University of Derby (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Derby Packed Lunch Trial
Record Dates: First submitted 2017-01-26; First posted 2017-04-07 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2017-01

CONDITIONS: Obesity, Childhood; Diet Modification
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: cluster randomised controlled trial
Who Masked: Participant
Masking Description: Parents and pupils will not be informed that their school is taking part in this research or that anonymous photographs will be taken of the contents of the lunch boxes brought into school by children in years 3 - 6.
  Written consent was obtained from the Head Teacher in all participating schools.
  Providing parents with information about the study is likely to change their behaviour and it will not be possible to assess whether the intervention itself has had an effect.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): No intervention materials will be distributed in the control schools during the intervention period.
- Intervention Group (Experimental): Intervention materials will be distributed to parents of children in years 3 - 6.
  Interventions: Behavioral: Behaviourally Informed Intervention Materials

INTERVENTIONS:
Behavioral: Behaviourally Informed Intervention Materials — The intervention consists of 7 separate components. The intervention components are to be delivered at three time-points (referred to as bundles). The bundles consist of:
  Bundle 1a - Letter to parents of children bringing a packed lunch to school, 'spot the difference' lunch box tag (attached to all lunchboxes) and a Handy Swaps Card.
  Bundle 1b - Letter to parents of children only having school meals and a Handy Swaps Card.
  Bundle 2 - Lunch box mixer with ideas for creating nutritious packed lunches. Bundle 3 - Shopping list, packed lunch planner and reward chart to support planning and monitoring progress.
  Arms: Intervention Group

SUMMARY:
Public Health England's (PHE) Behavioural Insights Team are leading and fully funding a randomised controlled research trial in collaboration with Derby City Council's Public Health Team and the Health and Social Care Research Centre at Derby University to test an intervention designed to help families provide healthier packed lunches for Primary School aged children.

DETAILED DESCRIPTION:
Children in Derby gain more weight during primary school than the national average. For 4-5 year olds, Derby is in the best performing quartile of English councils, with 20% having excess weight. However, by the age of 10-11 Derby drops to the second lowest quartile, with 35% of children having excess weight . In order to reduce childhood obesity in Derby, primary schools are a key area to focus on. Furthermore, it is a priority to focus on children living in deprived areas, as there is a strong relationship between deprivation and childhood obesity.

Research shows that packed lunches are higher in sugar, salt and saturated fat than school meals. , Furthermore, the nutritional gap between packed lunches and school meals has widened since the introduction of the food-based standards for school meals in 2006. A cross sectional survey, assessing packed lunches of 1,294 children in 87 primary schools, found only 1% met the standards for school meals in England, with 82% containing restricted snacks, i.e., crisps or confectionary, and 61% including sugar sweetened drinks. Therefore, significantly improving the quality of packed lunches could be an important step to reducing childhood obesity rates in Derby.

Previous research has highlighted that improving the quality of packed lunches can be challenging. For example, a UK-wide randomised controlled trial found that a "SMART lunch box" intervention had a positive impact on certain food groups but failed to reduce the overall calories in lunchboxes. The intervention, which included an extensive set of approaches, e.g., lunch bags, food boxes, wall charts, food games and stickers, increased vegetables packed by 11% and decreased savoury snacks packed by 14%, but failed to reduce confectionary and sweetened drinks . Other interventions, using educational videos and incentives aimed at children, had similar small, yet positive effects over a 12-month period . However, research has shown that relatively small, sustained behavioural changes can have a big cumulative impact: reducing calorie consumption by just 30-100 calories a day would have a considerable effect on obesity levels . The small effects of previous studies also highlight the importance of robustly evaluating any approach that is introduced.

In order to reduce childhood obesity in Derby, primary schools are a key area to focus on. Research shows that packed lunches are higher in sugar, salt and saturated fat than school meals, and a survey found only 1% of packed lunches met the standards for school meals in England . Therefore, significantly improving the quality of packed lunches could be an important step to reducing childhood obesity rates in Derby.

This trial is designed to test whether a multiple component intervention, focused on parents and developed with an understanding of the drivers behind behaviour, can increase the healthiness of packed lunches brought into school by reducing the presence of unhealthy items.

ELIGIBILITY:
Inclusion Criteria:

* All primary schools in Derby City
* Children in Years 3-6

Exclusion Criteria:

- Children in Years 1 - 2 due to universal provision of free school meals.

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2016-11-09 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
Proportion of lunchboxes that contain a sugary snack post-intervention | Data collected up to 6 months post intervention
  The proportion of lunchboxes that contain a sugary snack post-intervention
Proportion of lunchboxes that contain a chilled sugary dessert post-intervention | Data collected up to 6 months post intervention
  The proportion of lunchboxes that contain a chilled sugary dessert post-intervention

SECONDARY OUTCOMES:
Proportion of lunch boxes that contain any sugary food | Data collected up to 6 months post intervention
  The proportion of lunch boxes that contain any sugary food (i.e. either a sugary snack or chilled sugary dessert).
Total number of sugary food items | Data collected up to 6 months post intervention
  The total number of sugary food items (i.e. either a sugary snack or chilled sugary dessert)
Proportion of lunch boxes that contain crisps | Data collected up to 6 months post intervention
  The proportion of lunch boxes that contain crisps
Proportion of lunch boxes that contain a sugary drink | Data collected up to 6 months post intervention
  The proportion of lunch boxes that contain a sugary drink
Proportion of lunch boxes that contain fruit or vegetables | Data collected up to 6 months post intervention
  The proportion of lunch boxes that contain fruit or vegetables
The average nutritional value of sugary food items | Data collected up to 6 months post intervention
  The average nutritional value (e.g. grams of sugar, calories) of sugary food items

CONTACTS AND LOCATIONS:
Overall Officials: Tim Chadborn, PhD, Study Director — Public Health England; Amanda K Bunten, Doctorate, Principal Investigator — Public Health England
Locations (1):
- Amanda Bunten, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No